CLINICAL TRIAL: NCT02311465
Title: A Randomized Study of Early Palliative Care Integrated With Standard Oncology Care Versus Oncology Care Alone in Patients With Non-colorectal Gastrointestinal Malignancies.
Brief Title: A Randomized Study of Early Palliative Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Gordon Bernard, Professor of Medicine; Associate Vice-Chancellor for Research, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 141854
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Quality of Life
Keywords: Palliative Care
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palliative Care + Standard of Care (Experimental): Consenting patients will be approached by a research nurse to complete quality of life questionnaires (baseline measures) either in the oncology clinics or infusion clinics. Patients assigned to early palliative care will meet with a member of the palliative care team after enrollment and completion of the initial questionnaires to receive and review patient-oriented materials detailing palliative care services. Patients will then receive a comprehensive initial consult with a palliative care provider (a trained physician, nurse or nurse practitioner). Additional consults with the palliative care service will be scheduled approximately every 6 weeks for the duration of the study period (one year) at the discretion of the patient and palliative care provider.
  Interventions: Other: Palliative Care
- Standard of Care (No Intervention): Patients will receive standard care from their oncologist. An assessment of health related quality of life will be conducted at regular oncology clinic visits at baseline and 3,6,9,and 12 months.

INTERVENTIONS:
Other: Palliative Care — Components of the palliative care service intervention are expected to include:
  * Establishment of a palliative care plan
  * Care coordination by palliative care team
  * Informational, patient friendly materials supporting Palliative Care
  * Communication by palliative care team to all providers and teams involved in patient's care
  * Systematic collection of information, including identification of surrogate or health care proxy and advance care planning
  * Questionnaires capturing health related quality of life at regular intervals throughout the intervention period
  Other Names: Support Care
  Arms: Palliative Care + Standard of Care

SUMMARY:
The purpose of this research study is to find out whether it is better to introduce cancer patients to the palliative care team at a later date when there is a specific issue or problem or to introduce cancer patients to the palliative care team when first diagnosed before any specific issue or problem occurs.

DETAILED DESCRIPTION:
The investigators will conduct a one-year randomized, controlled study to evaluate the impact of an early, integrated palliative care services. The intervention will include comprehensive palliative care services delivered in conjunction with standard oncology care and patient friendly materials for high risk oncology patients. The investigators primary clinical endpoint will be health related quality of life, specifically focusing on measures of anxiety, depression, and well-being.

Secondary personalized palliative care outcomes are expected to include:

* Reduced deviations from care plan as captured in the medical record compared to the group who did not receive early, integrated palliative care services
* Reduced hospital utilization compared to the group who did not receive early, integrated palliative care services

ELIGIBILITY:
Inclusion Criteria:

* -Adults with newly diagnosed pancreatic, hepatocellular, esophageal, or stomach cancer
* Upcoming scheduled oncology clinic visit (2nd visit to the clinic) at Vanderbilt
* Ability to read and respond to questions in English
* Permission of oncology physician

Exclusion Criteria:

* -Receiving oncology care at non-Vanderbilt sites (to ensure appropriate follow-up)
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy: General (FACT-G) Health Related Quality of Life Questionnaire | 1 year
  The FACT Measurement System is a group of questions which measure health-related quality of life (QOL) in cancer patients. The FACT-G is a 26-item version that addresses multiple QOL dimensions including physical well-being, functional well-being, emotional well-being and social well-being. The response format of the FACT Measurement System consists of a 5-point Likert scale.

SECONDARY OUTCOMES:
PROMIS Depression Scale | 1 year
  Patient-Reported Outcome Measurement Information System (PROMIS) Depression scale is a highly reliable, validated, precise measures of patient-reported health status for physical, mental, and social well-being. The domains of depression are measured through four targeted questions each on a 5 point Likert scale.
PROMIS Anxiety Scale | 1 year
  Patient-Reported Outcome Measurement Information System (PROMIS) Anxiety scale is a highly reliable, validated, precise measures of patient-reported health status for physical, mental, and social well-being. The domains of anxiety are measured through four targeted questions each on a 5 point Likert scale.
Hospitalizations | 1 year
  Patient level data will be obtained for this study through retrospective chart review. Data to be collected from patients' charts include oncology medications and treatments, outcomes and interventions over the course of treatment (surgeries, adverse events, death), and hospitalizations. Clinical interventions, treatments, and events extracted from the charts will inform the investigators analyses regarding health care resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bernard, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States